CLINICAL TRIAL: NCT02261948
Title: Levosimendan Efficacy Assessment by Cardiopulmonary Exercise Test (CPET)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centro Cardiologico Monzino (Other)
Collaborators: Orion Corporation, Orion Pharma (Industry)
Responsible Party: Principal Investigator, Piergiuseppe Agostoni, Professor, Centro Cardiologico Monzino
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CCFM 199/312
Record Dates: First submitted 2014-07-22; First posted 2014-10-10 (Estimated); Results first posted 2015-11-06 (Estimated); Last update posted 2015-11-06 (Estimated); Status verified 2015-10

CONDITIONS: Heart Failure
Keywords: Cardiac Failure; Severe Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Simendan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Levosimendan (Active Comparator): Levosimendan must be diluted before the administration (500 ml of glucose). The intravenous infusion may be administered either by the peripheral or central. The dose and duration of therapy should be decided according to the patient's clinical condition and response to the drug. Treatment should be initiated with a loading dose of 6-12 mcg / kg infused over 10 minutes followed by a continuous infusion of 0.1 mcg / kg / min. A low infusion bolus (6 mcg / kg) is recommended for patients who have a concomitant intravenous treatment with vasodilators or inotropic. The patient's response should be evaluated during the infusion bolus or within 30 to 60 minutes and a dose adjustment based on clinical response.
  Interventions: Drug: Levosimendan
- Placebo (Placebo Comparator): Placebo must be diluted before the administration (500 ml of glucose). The intravenous infusion may' be administered either by the peripheral or central. The dose and duration of therapy should be decided according to the patient's clinical condition and response to the drug. Treatment should be initiated with a loading dose of 6-12 mcg / kg infused over 10 minutes followed by a continuous infusion of 0.1 mcg / kg / min. A low infusion bolus (6 mcg / kg) is recommended for patients who have a concomitant intravenous treatment with vasodilators or inotropic. The patient's response should be evaluated during the infusion bolus or within 30 to 60 minutes and a dose adjustment based on clinical response.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Levosimendan — Treatment should be initiated with a loading dose of 6-12 mcg / kg infused over 10 minutes followed by a continuous infusion of 0.1 mcg / kg / min.
  Other Names: SIMDAX
  Arms: Levosimendan
Drug: Placebo — Treatment should be initiated with a loading dose of 6-12 mcg / kg infused over 10 minutes followed by a continuous infusion of 0.1 mcg / kg / min.
  Arms: Placebo

SUMMARY:
The present study was conceived to evaluate the effects of levosimendan on cardiopulmonary exercise test (CPET) and DLCO ( Diffusion capacity of Lung for carbon monoxide) in patients with severe heart failure in stable clinical conditions (NYHA - New York Heart Association - class III, with a peak VO2 (Oxygen consumption ) < 12 ml/min/kg) on top of optimized standard therapy.

DETAILED DESCRIPTION:
Eligible patients should have chronic HF (Heart Failure -class NYHA III or IV) in stable clinical conditions. Inclusion criteria were: left ejection fraction (EF) at echocardiography ≤35%, age ≥18 years old, peak VO2 <12 ml/min/kg measured by a CPET, a standard optimized therapy for HF that include ACE-inhibitors, ARBs (angiotensin II Receptor Blocker), aldosterone blocking agents (spironolactone), diuretics, and beta-blockers.

The exclusion criteria are: ongoing mechanical ventilation; recent or acute coronary syndromes; sustained ventricular tachycardia or ventricular fibrillation; severe aortic or mitral regurgitation, or known malfunctioning artificial heart valve; uncorrected obstructive valvular disease; hypertrophic obstructive cardiomyopathy; uncorrected thyroid disease.

Patients will be randomly assigned by means of prepared letters to the levosimendan or placebo group stratified by clinical centre in a 1:1 allocation using block randomization. The placebo infusion will be coloured identically to its respective active counterpart. Patients and investigators will be kept blinded to the treatment allocation for the entire duration of the trial. Study drug will be infused with an injection speed between 6 and 20 ml/min based on blood pressure, without a bolus, for 24 hours.

Medical history, physical examination and a blood sample examination will be recorded: NYHA class, BNP (Brain Natriuretic Peptide), haemoglobin, creatinine, blood urea nitrogen (BUN) will be recorded before and 24 hours after the drug infusion.

A two-dimensional standard echocardiography evaluation will be performed at the admission in the hospital.

A maximal CPET performed on a cycle ergometer (Sensor Medics Ergo 800S and V-max, Yorba-Linda, CA) with a personalized ramp aimed at achieving peak exercise in 10 minutes will be performed before and 24 hours after the drug infusion. Expiratory O2, CO2 (Carbon dioxide) and ventilation (VE) will be measured breath by breath. Peak VO2 (Carbon dioxide production) was considered to be the highest VO2 achieved during the exercise. A 12-lead electrocardiogram will be also recorded. Spirometry and DLCO measurements will be performed before ad 24-hours after the drug infusion. . DLCO will be measured by the single breath-constant expiratory flow technique

ELIGIBILITY:
Inclusion Criteria:

* informed consent of the study signed
* severe heart failure in stable clinical condition (NYHA class III, peak VO2 <12 ml / kg / min) in optimized medical therapy. The clinical stability is defined by the stability of the therapy, the weight and urine output for 3 days

Exclusion Criteria:

* unstable patients from a clinical point of view, not in optimized therapy
* patients unable to perform a CPET (Cardiopulmonary Exercise Test) .
* are excluded from the protocol also patients with absolute contraindications to CPET (acute myocardial infarction, severe aortic stenosis, myocarditis or pericarditis, active, acute thromboembolism, sepsis,unstable angina, uncontrolled arrhythmia.
* age < 18 years.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2012-09; Primary Completion 2014-09 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Piergiuseppe Agostoni, MD, PhD, Principal Investigator — Centro Cardiologico Monzino,IRCCS
Locations (1):
- Centro Cardiologico Monzino, Milan, MI, Italy

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From September 2012 to December 2014 we enrolled forty-two patients who fulfilled the study inclusion/ exclusion criteria:19 patients received placebo and 23 received levosimendan. All patients was enrolled at Centro Cardiologico Monzino.
Pre-assignment Details: Eligible patients had advanced chronic heart failure and were admitted because of worsening HF (Heart Failure),although the patients included in the study had been returned to a stable clinical condition and were free from both inotrope support and other i.v. therapies for at least 48h prior to study inclusion, except for diuretics where needed.
Period: Overall Study
Arm/Group | Levosimendan | Placebo
Started | 23 | 19
Completed | 23 | 19
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Levosimendan | Placebo | Total
Number analyzed (Participants) | 23 | 19 | 42
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 4 | 10
  >=65 years | 17 | 15 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.39 (9.4) | 68.2 (8.3) | 69 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 7
  Male | 19 | 16 | 35
Region of Enrollment [Number; unit: participants]
  Italy | 23 | 19 | 42
NYHA class [Mean (Standard Deviation); unit: units on a scale] — New York Heart Association Class is the index used to classify the severity of symptoms referred by patients with heart failure. Lower index (1-2) is considered to have better outcome.
  units on a scale | 3.3 (0.4) | 3.2 (0.4) | 3.3 (0.47)

OUTCOME MEASURES:

1. Primary Outcome: Change in Peak VO2 (Oxygen Consumption )
Description: Primary endpoints: Levosimendan induced changes in peak VO2 (Oxygen consumption )
Time Frame: 48 hours
Measure: Mean (Standard Deviation); unit: ml/kg/min
Arm/Group | Levosimendan | Placebo
Number analyzed (Participants) | 23 | 19
ml/kg/min | 1.21 (1.9) | 0.48 (1.2)

2. Secondary Outcome: Changes in VE/VCO2
Description: Levosimendan induced changes on VE/VCO2 (VE: Expired Volume - VCO2: carbon dioxide production) relationship
Time Frame: 48 hours
Measure: Mean (Standard Deviation); unit: VE/VCO2 Slope
Arm/Group | Levosimendan | Placebo
Number analyzed (Participants) | 23 | 19
VE/VCO2 Slope | -5.34 (7) | -0.91 (4.7)

3. Secondary Outcome: Change in DLCO (Diffusion Lung CO)
Description: Levosimendan induced changes on DLCO ( Diffusion Lung CO). DLCO is measured by the single breath-constant expiratory flow technique (Sensor Medics 2200, Yorba Linda, CA) and we calculate also the DLCO adjusted for hemoglobin. Dilution of CH4 is used to measure alveolar volume.
Time Frame: 48 hours
Measure: Mean (Standard Deviation); unit: ml/mmHg/min
Arm/Group | Levosimendan | Placebo
Number analyzed (Participants) | 23 | 19
ml/mmHg/min | -0.96 (2) | 0.88 (3.14)

ADVERSE EVENTS:
Arm/Group | Levosimendan | Placebo
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/19
Other Adverse Events (participants affected / at risk) | 0/23 | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes